CLINICAL TRIAL: NCT00110435
Title: A Multicenter, Randomized, Double-blind, Parallel Group, 6-Week Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin Combination Tablet Versus Atorvastatin in Patients With Type 2 Diabetes Mellitus (T2DM) and Hypercholesterolemia
Brief Title: A Multicenter Study to Evaluate the Cholesterol Lowering Effects of Two Marketed Products in Patients With Type 2 Diabetes Mellitus and Hypercholesterolemia (MK-0653A-077)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-077; MK0653A-077; 2005_022
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes Mellitus; Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A, ezetimibe (+) simvastatin
Drug: Duration of Treatment: 4 wk placebo run in then 6 wk active
Drug: Comparator: atorvastatin

SUMMARY:
The purpose of this 10-week study is to compare the reduction in cholesterol following treatment with two different marketed drugs, in patients with type 2 diabetes mellitus and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 79 years who have a confirmed diagnosis of type 2 diabetes mellitus with elevated cholesterol levels may be eligible to participate in a study to assess the efficacy and safety of the two marketed drugs.

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Type 2 Diabetes Mellitus that is poorly controlled

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1229 (Actual)
Dates: Start 2005-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Percent reduction in LDL-C from baseline after 6 weeks of treatment

SECONDARY OUTCOMES:
Percent of patients attaining LDL-C <70 mg/dl after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Goldberg RB, Guyton JR, Mazzone T, Weinstock RS, Polis A, Edwards P, Tomassini JE, Tershakovec AM. Ezetimibe/simvastatin vs atorvastatin in patients with type 2 diabetes mellitus and hypercholesterolemia: the VYTAL study. Mayo Clin Proc. 2006 Dec;81(12):1579-88. doi: 10.4065/81.12.1579. PMID 17165637
- [Background] Tomassini JE, Mazzone T, Goldberg RB, Guyton JR, Weinstock RS, Polis A, Jensen E, Tershakovec AM. Effect of ezetimibe/simvastatin compared with atorvastatin on lipoprotein subclasses in patients with type 2 diabetes and hypercholesterolaemia. Diabetes Obes Metab. 2009 Sep;11(9):855-64. doi: 10.1111/j.1463-1326.2009.01061.x. Epub 2009 Jun 5. PMID 19508464